CLINICAL TRIAL: NCT02261558
Title: Effects of Clinical Music Improvisation on Resiliency in Adults Undergoing Infusion Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GCO 16-0838; 09-090 (Other: Beth Israel Medical Center)
Record Dates: First submitted 2014-07-24; First posted 2014-10-10 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clinical Improvisation Instrumental Music Therapy (Experimental): Clinical Music Therapy session, 20 minutes. Focus on instrumental improvisation
  Interventions: Other: Clinical Improvisation Instrumental Music Therapy
- Clinical Vocal Improvisation (Experimental): Clinical Music Therapy session, 20 minutes. Focus on vocal improvisation
  Interventions: Other: Clinical Vocal Improvisation
- Control Group (No Intervention): Participants enrolled in control group will complete the same study design, without having a clinical music improvisation

INTERVENTIONS:
Other: Clinical Improvisation Instrumental Music Therapy — Select an instrument of choice (and instruments for caregiver/s if applicable) Play/improvise and expand playing 10 minutes, inclusive of clinical improvisation (melody, harmony, timbre, and rhythmic idioms) where musical communication will be fostered and therapeutic goals will be addressed by the therapist in the music. Closure through verbal reflection and sharing (5 minutes)
  Arms: Clinical Improvisation Instrumental Music Therapy
Other: Clinical Vocal Improvisation — * 5 minutes of warm up. Select a few favorite songs of choice. Play/improvise and expand playing 10 minutes, inclusive of clinical improvisation (melody, harmony, timbre, and rhythmic idioms) where musical communication will be fostered and therapeutic goals will be addressed by the therapist in the music. Identify themes and issues addressed and/or paralleled in the song and/or within the self Closure through verbal reflection and sharing (5 minutes)
  Arms: Clinical Vocal Improvisation

SUMMARY:
This study will investigate the impact of music therapy on newly diagnosed patients with cancer undergoing chemotherapy. Measurements used at baseline, middle and end of first cycle will be the Resiliency Scale (Wagnild and Young 1993); The HADS scale (hospital anxiety depression scale, Zigmond and Snaith 1983 )and and The CAS scale for pain (Color Analysis Scale).

DETAILED DESCRIPTION:
The purpose of this research study is to examine clinical music therapy's impact on the resiliency of adults undergoing infusion therapy. This research study is being undertaken to learn about how creative music therapy modalities can affect the infusion therapy process. Infusion therapy often includes side effects which impact quality of life. Symptoms include pain, nausea and anxiety. For newly diagnosed patients anxiety accompanies adjustment to scheduling treatments and side effects. Typically patients receiving infusion therapy have no alternative focus for their mind and or body aside from the Infusion itself. Since the relationship between pain and anxiety is inter-related, altering one modality through a live music intervention may modify the impact of the other modality thus shifting the cycle and overall impact of pain and anxiety providing relief which leads to self soothing control measures. The current research will enroll patients newly diagnosed with either Lung, Breast, or Gastrointestinal Cancer that are treated in the Infusion Suite of SLRHC. 100 patients will be randomly assigned to three groups: clinical instrumental improvisation, clinical vocal improvisation or control. All enrolled participants will complete a survey which indicates their music preference, Resiliency Test , the Hospital Anxiety and Depression Scale (HADS), Visual Analogue Scale (VAS), and Body Pain Scale - Color Analysis Scale (CAS).

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* diagnosed with breast cancer, lung cancer, or gastro-intestinal cancer

Exclusion Criteria:

* Under 18
* past cancer(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2011-06; Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Resiliency Scale | At 6 months
  Research indicates that the majority of patients undergoing chemotherapy have extreme anxiety, particularly in the first round. . The music therapy implemented in the 2 treatment arms will be live and evaluated to meet the patients' culture, past medical history, past trauma upon assessment of psychological stressors. Resilience as measured through quantitative scale Wagnild, & Young (1993) that views daily activities and coping strategies that are often compromised with diseases that require frequent treatments.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | At 6 months
  The HADS provides entry and final treatment endurance in coping strategies related to anxiety and depression during disease treatment trajectories.
Music Psychotherapy Data Tool | At 6 months
  An informative questioner regarding the participant's musical preferences- favorite genres, artists or songs, and music history ( if applicable)- exposure to music through family members, and/or history of participation in a musical activity (such as social or private classes)
Visual Analogue Scale (VAS) | At 1 month
  The VAS is a single-item scale.A unidimensional measure of pain and stress intensity. A continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length, includes 5 levels of stress/pain (0,2,4,6,8,10), anchored by 2 verbal descriptors, one for each symptom extreme (no stress to worst possible stress).Tthe patient indicates the degree of stress he/she experiences by choosing one of the 5 levels on the scale. Respondents are asked to report "current" pain/stress intensity or "in the last 24 hours."
Visual Analogue Scale (VAS) | At 3 months
  The VAS is a single-item scale.A unidimensional measure of pain and stress intensity. A continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length, includes 5 levels of stress/pain (0,2,4,6,8,10), anchored by 2 verbal descriptors, one for each symptom extreme (no stress to worst possible stress).Tthe patient indicates the degree of stress he/she experiences by choosing one of the 5 levels on the scale. Respondents are asked to report "current" pain/stress intensity or "in the last 24 hours."
Visual Analogue Scale (VAS) | At 6 months
  The VAS is a single-item scale.A unidimensional measure of pain and stress intensity. A continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length, includes 5 levels of stress/pain (0,2,4,6,8,10), anchored by 2 verbal descriptors, one for each symptom extreme (no stress to worst possible stress).Tthe patient indicates the degree of stress he/she experiences by choosing one of the 5 levels on the scale. Respondents are asked to report "current" pain/stress intensity or "in the last 24 hours."
Body Pain Scale - Color Analysis Scale (CAS) | At 1 month
  An evaluative rating for pain, which offers the expression of pain through the patient's visual depiction, using crayon illustration on a sketch of a body figure . The participants are provided with a framed body figure, matched to their gender, including front and back of the body, in order for the participants to depict their pain experience with color.
Body Pain Scale - Color Analysis Scale (CAS) | At 3 months
  An evaluative rating for pain, which offers the expression of pain through the patient's visual depiction, using crayon illustration on a sketch of a body figure . The participants are provided with a framed body figure, matched to their gender, including front and back of the body, in order for the participants to depict their pain experience with color.
Body Pain Scale - Color Analysis Scale (CAS) | At 6 months
  An evaluative rating for pain, which offers the expression of pain through the patient's visual depiction, using crayon illustration on a sketch of a body figure . The participants are provided with a framed body figure, matched to their gender, including front and back of the body, in order for the participants to depict their pain experience with color.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Loewy, MT-BC, Principal Investigator — Mount Sinai Beth Israel
Locations (1):
- Beth Israel Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Bradt J, Dileo C, Myers-Coffman K, Biondo J. Music interventions for improving psychological and physical outcomes in people with cancer. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD006911. doi: 10.1002/14651858.CD006911.pub4. PMID 34637527
- [Derived] Mondanaro JF, Sara GA, Thachil R, Pranjic M, Rossetti A, EunHye Sim G, Canga B, Harrison IB, Loewy JV. The Effects of Clinical Music Therapy on Resiliency in Adults Undergoing Infusion: A Randomized, Controlled Trial. J Pain Symptom Manage. 2021 Jun;61(6):1099-1108. doi: 10.1016/j.jpainsymman.2020.10.032. Epub 2020 Nov 2. PMID 33152443